CLINICAL TRIAL: NCT04315805
Title: Integrative Yoga Therapy for Patients With Chronic Pain and Psychological Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU07
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain; Psychological Distress
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Yoga Therapy (Experimental): Integrative Yoga Therapy will be provided by yoga therapist once a week and participants will be encouraged to practice at home once or twice a day.
  Interventions: Other: Integrative Yoga Therapy
- Wait-list Control (No Intervention): Participants in waiting list will serve as control group for the intervention period. After the ftherapy group has received treatment, the same program will be offered to participants in the wait-list control group.

INTERVENTIONS:
Other: Integrative Yoga Therapy — Yoga therapy will be based on personalised care consisting of Yoga relaxing posture, strengthening exercise, Yoga breathing, meditative psychotherapy, sound and imagery yoga practices, relaxation, yoga diet and life style management.
  Arms: Integrative Yoga Therapy

SUMMARY:
This study will be a randomized wait list controlled trial studying the efficacy of an Integrative Yoga Therapy for patients with chronic pain and psychological distress. Individualised yoga program will consist of a 8-week guided self-help program.

This study will primarily investigate whether an individually tailored yoga can be beneficial for patients suffering from chronic pain reducing pain, anxiety depression, while improving overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Experienced pain for > 3 months
* Experiences at least one type of psychological distress such as: depression, anxiety, insomnia or stress
* Willing to provide informed consent

Exclusion Criteria:

* Severe medical or psychiatric conditions
* Alcohol or substance abuse
* Active suicidality
* Terminal illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain Severity: Visual Analogue Scale | From baseline to 8-week post intervention
  Visual Analogue Scale ranging between 0-10 where 0 is no pain at all and 10 is worst pain
Pain Disability | From baseline to 8-week post intervention
  Change in pain disability using Pain Disability Index (PDI) with 7 item.Each item scores on 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability
Symptoms of depression and anxiety | From baseline to 8-week post intervention
  Hospital Anxiety Depression Scale with 14 item. Each item on the questionnaire is scored from 0-3 where higher score represents increased anxiety and depression levels

SECONDARY OUTCOMES:
Insomnia symptoms | From baseline to 8-week post intervention
  Insomnia Severity Index has seven questions each scores between 0-4. Higher score defines severity of clinical insomnia
Mental well-being | From baseline to 8-week post intervention
  The Short Warwick-Edinburgh Mental Wellbeing Scale; Minimum score: 7; maximum score: 35; higher score indicates greater level of wellbeing
Self Efficacy: Pain Self-Efficacy Questionnaire (PSEQ)- 2 item scale | From baseline to 8-week post intervention
  Pain Self-Efficacy Questionnaire (PSEQ)- 2 item scale

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK
Locations (1):
- Karyalaya, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided